CLINICAL TRIAL: NCT04991792
Title: Evaluation of the Effect of an Infant Formula Containing Synbiotics on the Composition of the Gut Microbiota in Infants Born Via Caesarean Section
Brief Title: Effect of an Infant Formula With Synbiotics in Infants Born Via Caesarean Section
Acronym: GOLF-CS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HiPP GmbH & Co. Vertrieb KG (Industry)
Collaborators: University Multiprofile Hospital for Active Treatment Dr. Georgi Stranski EAD, Pleven, Bulgaria (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 510646
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Gut Microbiota
Keywords: Caesarean Section; Microbiota; Infant Formula; Infants
MeSH Terms: interventions — Synbiotics; Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Standard Infant Formula with synbiotics (CS-born) (Experimental): CS born infants, randomized to receive infant formula with synbiotics
  Interventions: Other: Intervention Group 1: Infant Formula with synbiotics
- Standard Infant Formula with prebiotics (CS-born) (Experimental): CS born infants, randomized to receive infant formula with prebiotics
  Interventions: Other: Intervention Group 2: Infant Formula with prebiotics
- Control Group 1: Standard Infant Formula (CS-born) (Active Comparator): CS born infants, randomized to receive standard infant formula without synbiotics
  Interventions: Other: Control Group 1 and 2: Infant Formula without synbiotics
- Control Group 2 : Standard Infant Formula (VD-born) (Active Comparator): VD born infants, receiving standard infant formula without synbiotics (self-selected for formula-feeding = non-randomized)
  Interventions: Other: Control Group 1 and 2: Infant Formula without synbiotics
- Reference Group 1: Breastfed (CS-born) (No Intervention): CS-born infants, receiving exclusive breast-feeding with mother's own breast milk (non-randomized)
- Reference Group 2: Breastfed (VD-born) (No Intervention): VD-born infants, receiving exclusive breast-feeding with mother's own breast milk (non-randomized)

INTERVENTIONS:
Other: Intervention Group 1: Infant Formula with synbiotics — Infants will receive infant formula during the first 6 months of life
  Arms: Standard Infant Formula with synbiotics (CS-born)
Other: Intervention Group 2: Infant Formula with prebiotics — Infants will receive infant formula during the first 6 months of life
  Arms: Standard Infant Formula with prebiotics (CS-born)
Other: Control Group 1 and 2: Infant Formula without synbiotics — Infants will receive infant formula during the first 6 months of life
  Arms: Control Group 1: Standard Infant Formula (CS-born); Control Group 2 : Standard Infant Formula (VD-born)

SUMMARY:
A multi-centre, randomized, parallel-group, double-blind, controlled, exploratory clinical trial is conducted to assess the positive effect of feeding a formula containing synbiotics (pre- and probiotics) on the composition of the gut microbiota in caesarean section (CS) born healthy term infants within the first 6 months of life.

DETAILED DESCRIPTION:
Since caesarean section (CS)-born infants show dysbiotic microbial colonization during the first weeks of life, exclusive breastfeeding is the feeding mode of choice for these infants. However, since CS births are often associated with breast-feeding difficulties, it is of importance to feed an microbiota-supportive infant formula. This study is designed to investigate whether an infant formula supplemented with synbiotics positively affects the microbial composition, gastrointestinal characteristics and the proper function of the immune system in CS-born infants, compared to feeding a standard infant formula without synbiotics in either CS- and vaginal-born infants during the first 6 months of life. The growth of the infants as well as tolerance, infectious diseases and allergies will also be assessed. In order to investigate the effect of different birth modes and feeding conditions on the microbiota, the study population will include healthy term infants, born either by CS or by VD, additional groups receive human milk or formula with prebiotics only. Additionally, if the parents agree, their infant will be followed up until 24 months of age with a special focus on the prevention of infections and allergies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants
* Female or male gender
* Gestational age ≥37 weeks, <42 weeks
* Singleton, born by caesarean section or vaginally born
* Birth weight between ≥2500g and ≤4200g with a regular weight gain without any signs of developmental delays or growth disorders according to investigator opinion
* Uncomplicated early course of neonatal period
* Age at enrolment: 5 +/-1 days of life
* Infants whose parent(s)/ legal authorized representatives (LAR(s)) have reached the legal age of majority in Bulgaria
* Infants whose parent(s)/ LAR(s) are capable of and willing to comply with the protocol and have signed the informed consent form in accordance with legal requirements
* At least one of the legal representatives is affiliated to a health security/insurance or equally
* Infants whose parent(s)/ LAR(s) are willing to comply with the feeding regimen during the intervention period. Infant's parent(s)/ LAR(s) will decide which feeding regimen will be used (infant formula or breast milk)
* Parents/ LARs who agree to not use any sort of other formula than provided during the study

Exclusion Criteria:

* Intensive care prior to or at Baseline Visit
* UV-treatment of jaundice and clinical significant jaundice prior to Baseline Visit (according to investigator opinion)
* Known immune deficiency
* Serious acquired or congenital diseases, chromosomal anomalies (if known)
* Serious pre-natal and/or serious post-natal disease before enrolment (per investigator's medical diagnosis)
* Infants or mothers under antibiotic treatment before Baseline Visit (only for vaginally born and breastfed infants) or at Baseline Visit (all groups)
* Infants requiring infant formula intake other than those specified in the protocol (formula for special medical purposes (FSMP), formula with hydrolyzed protein (allergy risk)
* Infant's supplementation or formula intake, which contains probiotics, prebiotics, dietary fibres or synbiotics before and during study
* Feeding difficulties or formula intolerance according to investigator's opinion
* Currently participating or having participated in another clinical trial since birth
* Reason to presume that the infant's parent(s)/LAR(s) are unable to meet the study plan requirements, such as drug/alcohol abuse, psychological or linguistic incapability, chronic or mental diseases
* Infants born to mothers with medical conditions that require prescription medication (coagulation abnormalities, if acetylsalicylic acid was not stopped at 35 weeks GA according to guidelines, mothers treated with Methyldopa, ACE inhibitors, breastfeeding mothers treated with L-thyroxine, diabetic mothers, epileptic mothers)
* Any smoking, drug or alcohol intake by the mother during the last two trimesters of pregnancy
* Mother's weight gain >18 kg during pregnancy

Ages: 4 Days to 6 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 486 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2024-07-07 (Actual)

PRIMARY OUTCOMES:
Assessment whether an infant formula containing synbiotics positively affects the composition of the gut microbiota in CS-born infants compared to a standard formula (without synbiotics) or breast-feeding within the first 6 months of life | 6 months duration

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Assoc. Prof. Dr. Atanasova, MD, PhD, Principal Investigator — "Dr. Georgi Stranski" EAD, 91 "Vladimir Vazov" Str., 5809 Pleven, Bulgaria
Locations (1):
- University multiprofile hospital for active treatment "Dr. Georgi Stranski" EAD, Pleven, Bulgaria

IPD SHARING:
Plan to Share IPD: Undecided